CLINICAL TRIAL: NCT04606914
Title: Single-Arm Phase II Study of Carboplatin and Mirvetuximab Soravtansine in First-Line Treatment of Patients Receiving Neoadjuvant Chemotherapy With Advanced-Stage Ovarian, Fallopian Tube or Primary Peritoneal Cancer Who Are Folate Receptor α Positive
Brief Title: Study of Carboplatin and Mirvetuximab Soravtansine in First-Line Treatment of Patients Receiving Neoadjuvant Chemotherapy With Advanced-Stage Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rebecca Arend, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300005764
Record Dates: First submitted 2020-10-16; First posted 2020-10-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer; Fallopian Tube; Primary Peritoneal Cancer
Keywords: First line treatment; Advanced epithelial ovarian cancer; mirvetuximab soravtansine; IMGN853
MeSH Terms: conditions — Ovarian Neoplasms | interventions — mirvetuximab soravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: alpha receptor positive_neoadjuvant chemotherapy regimen (Experimental): * IV Carboplatin AUC 5 (Q21 days) 7 cycles (first cycle is Carbo alone, dosing for C1D1 will be provider's choice)
  * IV Mirvetuximab 6 mg/kg (adjusted ideal body weight) day 1 (Q21 days) 6 cycles (starting with cycle #2)
  Interventions: Drug: mirvetuximab soravtansine (MIRV; IMGN853)
- Arm B: alpha receptor negative (No Intervention): If a patient is found to be negative for FRα expression, they will be ineligible to receive the study treatment under the main study (Arm A). FRα negative patients will be enrolled under the biomarker-only arm (Arm B), and their treating physician can select the treatment they deem appropriate.

INTERVENTIONS:
Drug: mirvetuximab soravtansine (MIRV; IMGN853) — Mirvetuximab soravtansine (also known as IMGN853 and MIRV) is an antibody-drug conjugate (ADC) that consists of a high affinity humanized monoclonal antibody against folate receptor α (FRα, the protein product of the folate receptor 1 [FOLR1] gene) that is conjugated to a cytotoxic maytansinoid by the hindered disulfide succinimidyl 4-(pyridin-2-yl)disulfanyl)-2-sulfo-butyrate linker (sulfo-SPDB) linker. FRα is a glycosyl-phosphatidylinositol (GPI)-linked protein, which shows limited normal tissue expression and high expression on the surface of solid tumors, particularly epithelial ovarian cancer, fallopian tube cancer, and primary peritoneal cancer (referenced herein collectively as EOC), endometrial cancer, non-small cell lung cancer (NSCLC), and renal cell cancer.
  Arms: Arm A: alpha receptor positive_neoadjuvant chemotherapy regimen

SUMMARY:
The proposed study design is a single arm Phase II trial to document the feasibility of carboplatin-mirvetuximab - in patients with advanced-stage EOC. Patients with biopsy confirmed, newly diagnosed, advanced-stage serous EOC deemed appropriate for NACT will have their tumors evaluated for FRα receptor over-expression via a centralized immunohistochemical assay (IHC) and identified as appropriate for study participation if IHC staining is PS2+ in >75% of cells (40% of all serous patients). Eligible patients will receive NACT with one cycle of carboplatin, followed by mirvetuximab + carboplatin (if FRα +) every 21 days for three cycles prior to interval cytoreductive surgery (iCRS). A total of 70 will be included in the study. Following completion of 4 cycles total of NACT and after allowing for appropriate recovery of cycle # 4, patients eligible for surgery, will undergo an iCRS. Patients will then complete 3 more cycles of mirvetuximab + carboplatin for a total of 7 intended cycles of treatment. It is up to the treating physician if they want to add bevacizumab to the last 2 cycles or use any type of maintenance therapy. The decision to add bevacizumab or use maintenance therapy does not need to be made upfront. Patients will sign a screening consent form prior to tissue biopsy. If a patient is found to be FRα negative, their treating physician can select the treatment they deem appropriate and the patient will be declared a screen failure. Patients with BRCA mutations are not excluded from this trial and are allowed to receive standard of care maintenance therapy including bevacizumab and/or PARP inhibitors.

DETAILED DESCRIPTION:
Mirvetuximab soravtansine (also known as IMGN853 and MIRV) is an antibody-drug conjugate (ADC) that consists of a high affinity humanized monoclonal antibody against folate receptor α (FRα, the protein product of the folate receptor 1 [FOLR1] gene) that is conjugated to a cytotoxic maytansinoid by the hindered disulfide succinimidyl 4-(pyridin-2-yl)disulfanyl)-2-sulfo-butyrate linker (sulfo-SPDB) linker. FRα is a glycosyl-phosphatidylinositol (GPI)-linked protein, which shows limited normal tissue expression and high expression on the surface of solid tumors, particularly epithelial ovarian cancer, fallopian tube cancer, and primary peritoneal cancer (referenced herein collectively as EOC), endometrial cancer, non-small cell lung cancer (NSCLC), and renal cell cancer. The selective upregulation of FRα in solid tumors and the potent and selective cytotoxicity of MIRV against FRα-positive tumor cells demonstrated in nonclinical studies and clinical studies to date provide rationale for further investigation of MIRV in the treatment of FRα-positive tumors.

Ovarian cancer is a lethal disease with 22,530 new cases and 13,980 deaths expected in 2019 in the US. The estimated number of new EOC cases in the EU (EU27) in 2012 was 44,149 with 29,758 deaths. The overall 5-year survival for EOC patients is only 44%. Besides the incorporation of a platinum- and taxane-based chemotherapy regimen into the upfront treatment, no major strides have been made to improve overall survival (OS) following EOC diagnosis.

Standard of care chemotherapy includes every 21-day paclitaxel and carboplatin, weekly paclitaxel and every 21-day carboplatin. Recently, bevacizumab was approved to be given with and to follow intravenous chemotherapy in front line ovarian cancer based on the PFS advantage demonstrated in GOG 218 and ICON7. This study continued bevacizumab for 15 cycles post completion of 6 cycles of chemotherapy. In evaluating the morphology of the Kaplan Meier curves from both these trials, it is apparent that there is an inflexion in the curves at the point where the bevacizumab is discontinued. To evaluate whether further continuation of bevacizumab would improve PFS, AGO-OVAR17 (BOOST study) is evaluating 15 versus 30 cycles of bevacizumab following front line chemotherapy. These results are anticipated in 2021. Given the above data, this trial as designed, will not include a specific maintenance portion, but physicians can choice what type of maintenance therapy, if any, they give at the completion of at least 7 cycles of platinum +Mirvetuximab soravtansine.

Despite considerable improvements in primary therapy, 80% of the patients with advanced EOC are expected to relapse during or after treatment with platinum-containing regimens. Disease recurring within 6 months of platinum-based chemotherapy is classified as platinum resistant, whereas, disease recurring longer than 6 months after therapy is termed platinum sensitive.

Those patients with PROC who have received prior bevacizumab, either in the platinum-resistant or in the platinum-sensitive setting, have few options. They typically receive subsequent single-agent chemotherapy. Unfortunately, response rates to single-agent chemotherapy are modest (~10 to 15%) and DOR is typically 4 to 8 months. Similarly, OS is poor (median ~11 to 14 months). Because PROC remains a significant unmet medical need, the National Comprehensive Cancer Network (NCCN) guidelines recommend that platinum-resistant patients participate in clinical trials.

The proposed neoadjuvant chemotherapy regimen is as follows:

IV Carboplatin AUC 5 day 1 (Q21 days) 7 cycles (first cycle is Carbo alone) IV Mirvetuximab 6 mg/kg (adjusted ideal body weight) day 1 (Q21 days) 6 cycles (starting with cycle #2)

Patients will continue to receive MIRV until they present with PD per RECIST 1.1, as assessed by study Investigator, unacceptable toxicity, withdraw consent, or death, whichever comes first, or until the Sponsor terminates the study. Study treatment and/or participation in the study may be discontinued at any time at the discretion of the Investigator. The following may be reasons for the Investigator to remove a patient from the study drug:

The patient suffers an intolerable Adverse Event (AE). Noncompliance, including failure to appear at one or more study visits Study treatment and/or participation in the study may be discontinued at any time at the discretion of the Investigator.

The reason for treatment discontinuation must be captured in the clinical trial database. Any AEs experienced up to the point of discontinuation and 30 days thereafter must be documented. All serious adverse events (SAEs), and those AEs assessed by the Investigator as at least possibly related to study drug should continue to be followed until they resolve or stabilize, whichever comes first. Patients will continue to be followed for OS, after discontinuing study drug.

For purposes of this study, the period of safety observation extends from the time of informed consent until the 30-Day Follow-up visit unless additional follow-up safety information is requested as described in Section 9.3. Short-term follow-up for patients who discontinue study drug without documented PD will be followed per RECIST 1.1 every 12±1 weeks until PD, until the patient starts new anticancer treatment, the patient dies, or the patient withdraws consent, whichever comes first. All patients will be followed every 3±1 months for survival until death, lost to follow-up, withdrawal of consent for survival or until EOS, whichever comes first.

Radiographic tumor evaluation by CT or MRI of chest, abdomen, and pelvis will be performed within 28 days before first dose of study drug, before IDS within 21 days after C4D1, and a minimum of 21 days following C7D1. The same method of radiologic assessment used at Screening must be used at all subsequent radiographic evaluations.

Tumor response will be assessed by the Investigator using RECIST v1.1. Response as determined by the Investigator will be recorded in the clinical trial database.

The sample size will comprise of approximately 70 patients from the University of Alabama at Birmingham.

The primary objective will be feasibility (the proportion of consented patients who successfully obtain biopsy confirmation of disease status and IHC analysis of FRα receptor status prior to starting treatment with mirv). The primary analysis will include all consenting patients. Patients who obtain both the biopsy confirm and are FRα positive will be considered feasibility successes. The remainder of the consenting sample will be considered feasibility failures, regardless of the reason for failure.

Key Secondary Objective will be progression free survival (PFS), percentage disease free at 2 years, ORR prior to interval debulking surgery (IDS) per iRECIST 1.1 and GCIG CA-125 criteria, and percentage of optimal cytoreduction and pathological complete response (PCR) at IDS.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy-confirmed high grade serous epithelial ovarian cancer.
* Patients must present with stage III or IV disease and be appropriate to receive neoadjuvant chemotherapy
* Patients must be willing to provide an archival tumor tissue block or slides, or undergo procedure to obtain a new biopsy using a low-risk, medically routine procedure for immunohistochemistry (IHC) confirmation of FRα positivity
* Patients must have a performance status of 0 or 1.
* Patient's tumor must be positive for FRα expression as defined by a score of PS2+ intensity in >75% of cells
* Patients must have adequate hematologic, liver and kidney functions defined as:
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (1,500/μL)
* Platelet count ≥ 100 x 109/L (100,000/μL) without platelet transfusion in the prior 10 days
* Hemoglobin ≥ 9.0 g/dL
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x ULN
* Serum bilirubin ≤ 1.5 x ULN (patients with documented diagnosis of Gilbert syndrome are eligible if total bilirubin < 3.0 x ULN)
* Serum albumin ≥ 2 g/dL
* Patients must be willing and able to sign the informed consent form (ICF) and to adhere to the protocol requirements
* Women of childbearing potential (WCBP) must agree to use highly effective contraceptive method(s) (as defined in Section 5.8.6 while on MIRV and for at least 4 months after the last dose
* WCBP must have a negative pregnancy test within the 4 days prior to the first dose of MIRV

Exclusion Criteria:

* Patients who have previously been treated with a systemic anti-cancer therapy
* Patients with low-grade serous, endometrioid, clear cell, or mucinous histology
* Patients with active or chronic corneal disorders, history of corneal transplantation, or active ocular conditions requiring ongoing treatment/monitoring, such as uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema, and /or monocular vision
* Patients with serious concurrent illness or clinically relevant active infection, including, but not limited to the following:
* History of hepatitis B or C infection (whether or not on active antiviral therapy)
* History of human immunodeficiency virus (HIV) infection
* Any other concurrent infectious disease requiring IV antibiotics within 2 weeks prior to the first dose of MIRV
* Patients with a history of multiple sclerosis (MS) or other demyelinating disease and/or Lambert-Eaton syndrome (paraneoplastic syndrome)
* Patients with clinically significant cardiac disease including, but not limited to, any of the following:
* Myocardial infarction ≤ 6 months prior to first dose
* Unstable angina pectoris
* Uncontrolled congestive heart failure (New York Heart Association > class II)
* Uncontrolled ≥ Grade 3 hypertension (per CTCAE)
* Uncontrolled cardiac arrhythmias
* Patients with a history of hemorrhagic or ischemic stroke within 6 months prior to enrollment
* Patients with a history of cirrhotic liver disease (Child-Pugh Class B or C)
* Patients with a previous clinical diagnosis of noninfectious interstitial lung disease (ILD), including noninfectious pneumonitis
* Patients requiring use of folate-containing supplements (eg, folate deficiency)
* Patients with prior hypersensitivity to monoclonal antibodies (mAb)
* Women who are pregnant or breastfeeding
* Patients who received prior treatment with MIRV or other FRα-targeting agents
* Patients with untreated or symptomatic central nervous system (CNS) metastases
* Patients with a history of other malignancy within 3 years prior to enrollment Note: patients with tumors with a negligible risk for metastasis or death (eg, adequately controlled basal-cell carcinoma or squamous-cell carcinoma of the skin, or carcinoma in situ of the cervix or breast) are eligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with biopsy-confirmed high grade serous epithelial ovarian cancer
Enrollment: 70 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | Baseline through 2 years
  To assess percentage of patients with advanced-stage ovarian, fallopian tube, and peritoneal cancers per Response Evaluation Criteria in Solid Tumors (RECIST)1.1 and Gynecological Cancer Intergroup Cancer antigen 125 (GCIG CA-125) criteria.
Objective response rate (ORR) | Baseline through 2 years
  To assess ORR per iRECIST 1.1 and GCIG CA-125 criteria
Radiographic tumor assessment per RECIST v1.1 criteria | Baseline through 2 years
  Radiographic tumor response by CT or MRI of chest, abdomen, and pelvis using RECIST v1.1

SECONDARY OUTCOMES:
Serum Cancer Antigen 125 (CA-125) assessments | Baseline through 2 years
  Serum CA-125 will be assessed by the same laboratory throughout the study.
Safety profile of treatment with carboplatin-mirvetuximab soravtansine according to CTCAE v4.03 | Baseline through 2 years
  To determine the nature and degree of toxicity oftreatment with carboplatin-mirvetuximab soravtansine according to Common Terminology Criteria for Adverse Events (CTCAE) v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Arend, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (9):
- United States (9):
  - University of Alabama at Birmingham Womens & Infants Center, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - University of Minnesota - Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Oxford, Mississippi
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - University of Virginia, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No